CLINICAL TRIAL: NCT02510521
Title: Effects of Neuro-myo-electrical Stimulation on Insulin Sensitivity in Patients With Type 2 Diabetes
Acronym: ELECTRODIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-063
Record Dates: First submitted 2015-07-23; First posted 2015-07-29 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- in rest situation (Placebo Comparator): No intervention during one week. Daily usual activities are allowed.
  Interventions: Other: rest situation
- after acute muscle exercise by NMES (Experimental): A working session of 20 minutes with three sequences electrostimulation:
  * warming-up sequence
  * work sequence (starting at 50% of the intensity achieved during warm-up)
  * relaxation sequence
  Electrostimulation relates both quadriceps are stimulated simultaneously and jointly. During the sessions, the patient sits on a chair or on a chair, legs bent at 90 °. So that there is no extension of the legs when electrostimulation (which could be painful), a strap is placed behind the legs of the chair or armchair and holds the pegs.
  Interventions: Device: acute muscle exercise by NMES
- after a daily workout sequence with NMES in one week (Experimental): Working sessions of 20 minutes 7 days in a row, including :
  * warming-up sequence
  * work sequence (starting at 50% of the intensity achieved during warm-up)
  * relaxation sequence
  Electrostimulation relates both quadriceps are stimulated simultaneously and jointly. During the sessions, the patient sits on a chair or on a chair, legs bent at 90 °. So that there is no extension of the legs when electrostimulation (which could be painful), a strap is placed behind the legs of the chair or armchair and holds the pegs.
  Interventions: Device: daily workout sequence with NMES in one week

INTERVENTIONS:
Device: acute muscle exercise by NMES
  Arms: after acute muscle exercise by NMES
Device: daily workout sequence with NMES in one week
  Arms: after a daily workout sequence with NMES in one week
Other: rest situation
  Arms: in rest situation

SUMMARY:
Type 2 diabetes is a major public health problem because of its increasing prevalence and morbidity and mortality that accompanies it. Therapeutic management of this pathology, lifestyle measures, dietary and physical activity are fundamental. Their observance is unfortunately too often insufficient, leading to a therapeutic climbing with first oral antidiabetic (OAD) then the use of insulin therapy.

Yet there is now ample evidence that physical activity improves glucose control in these patients in particular improving insulin sensitivity after a training period but also after a single session of physical activity.

Neuro-myo-electrical stimulation (NMES) is used in common clinical practice in physical therapy, patients with neurological or after orthopedic surgery in particular. In fact, this method enables improvement of volume and strength, even for denervated muscles. Recent studies have also shown the benefits of NMES in situations of cardiac or respiratory readjustments. In addition, NMES is used by top athletes supplements classical training in order to develop muscle strength or speed recovery.

Investigators propose to test the impact of bilateral quadriceps NMES on insulin sensitivity in type 2 diabetic patients treated with OAD (excluding glitazone). To do this, investigators plan to assess their insulin sensitivity by the reference method of hyperinsulinemic euglycemic clamp before surgery, after a single session of bilateral quadriceps NMES and after a sequence of daily training 6 days a quadriceps NMES bilateral.

Investigators hope to show an improvement in insulin sensitivity by this method, which would constitute an alternative to physical activity in the treatment of diabetes type 2. This procedure would be particularly interesting in diabetic subjects with type 2 counter- indications or an inability to perform a conventional physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-75 years of age:
* Type 2 diabetes,
* in a context of overweight BMI upper than 25 kg / m²,
* a glycated hemoglobin included between 6 and 9%,
* treated with oral antidiabetic (non glitazone) and / or GLP1 analogs (stable treatment for 3 months).
* Patient who signed informed consent.

Exclusion Criteria:

* Type 1 diabetes
* Children or adolescents under 18 years.
* Patients over 75 years.
* Pregnancy.
* Patient intense practicing regular physical activity and do not wish to interrupt the time of the study
* Patients with painful joint disease of the knee mobilization (osteoarthritis, inflammatory arthritis), any severe neuromuscular disease (diabetic neuropathy with pain, cramps, paresthesia, hypoesthesia, degenerative muscle disease).
* Patients with unstable ischemic heart disease or arterial disease severe lower limbs.
* Presence of a pacemaker (pacemaker).
* Epilepsy
* Patients insulin applicants
* Treatment with glitazone.
* Sepsis or other intercurrent acute disease (heart attack, angina ..).
* Patients with skin lesions of any kind (wounds, inflammations, burns, irritations, eczema, etc.) nearby with areas for electrodes NMES
* Patients unable to comply with the safety instructions of the NMES device at home
* Patient unable to submit to medical monitoring study for geographical, social or psychological.
* Patients under guardianship or trusteeship.
* Patient included in another biomedical research protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity measured by the reference euglycemic hyperinsulinemic clamp technique | change over time : baseline, week 1, end of week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology Unit and Clinical Research Center Basse Normandie, University Hospital of Caen, Caen, France